CLINICAL TRIAL: NCT01879215
Title: Patella Femoral Changes Following Tibial Nailing: Does Approach Matter?
Brief Title: T1Rho MRI Evaluation of Patellofemoral Changes After Tibial IM Nailing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 817841
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Acute Tibial Fracture Requiring Intramedullary Nailing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suprapatellar Approach (Active Comparator): Suprapatellar Approach to Intramedullary Nailing. Surgeons will be allowed to use any size intramedullary tibial nail through an suprapatellar incision and splitting the quadriceps tendon.
  Interventions: Procedure: Intramedullary nailing of the tibia
- Infrapatellar Approach (Active Comparator): Infrapatellar Approach Intramedullary Nailing. Surgeons will be allowed to use any size intramedullary tibial nail through an infrapatellar incision using either a medial parapatellar approach or a transpatellar approach. The knee will then be scanned using T1Rho MRI at 2 weeks postoperatively and 6 months postoperatively.
  Interventions: Procedure: Intramedullary nailing of the tibia

INTERVENTIONS:
Procedure: Intramedullary nailing of the tibia — Standard care surgery

SUMMARY:
This study will utilize T1-Rho MRI to evaluate the effect of intramedullary nailing on patellofemoral articular cartilage when the surgery is performed using the infrapatellar vs. the suprapatellar approach. Subjects will be randomized to one or the other standard care surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated tibial shaft fractures indicated for intramedullary nailing,
2. Acute tibia fractures,
3. Closed or open tibia fractures,
4. Skeletally mature patient between the ages of 21 and 50,
5. No prior history of knee surgery,
6. No prior history of knee pain,
7. No history of degenerative joint disease or inflammatory arthropathy
8. Not pregnant or known to be under the jurisdiction of the Department of Corrections
9. Able to provide informed consent.
10. Qualifies for standard care tibial IM nailing using either a suprapatellar or infrapatellar approach with no physician preference or definitive clinical indication for one or the other approach
11. Ability to communicate, read, and write in English
12. Intent of subject to receive follow up fracture care at the PI's institution.

Exclusion Criteria:

1. Tibial fractures requiring articular reconstruction (tibial plateau fractures and pilon fractures),
2. Periprosthetic fractures,
3. Nonunions or malunions,
4. History of previous knee surgery,
5. History of preexisting knee pain,
6. History of degenerative arthritis or inflammatory arthropathy, any evidence of degenerative changes of pre-operative knee radiographs, and any concomitant injury to that limb.
7. Any contraindication to MRI imaging
8. Retained stainless steel hardware proximal to the knee joint including, but not limited to prior knee replacement.
9. Under age 18 at the time of presentation, pregnant or planning to become pregnant within the study period, or under the jurisdiction of the Department of Corrections.
10. Inability to provide informed consent
11. Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study
12. Insurance or other circumstantial restriction that would prohibit or interfere with the subject's ability to receive follow up care at the PI's institution.
13. Any condition, acute or chronic, that in the opinion of the attending physician or the Principal Investigator, would contraindicate participation in this study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2020-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
T1Rho MRI to quantify patellofemoral cartilage changes after IM nailing of the tibia as a primary treatment for acute tibial fractures. | Up to 6 months post-discharge
  The difference in proteoglycan content of patellofemoral articular cartilage as quantified using spin lattice relaxation in a rotating frame (T1ρ MRI weighted image) at 6 months post-hospital discharge between two groups randomized to undergo either a suprapatellar or infrapatellar approach to tibial IM nailing.

SECONDARY OUTCOMES:
SF-36 | Pre-op, 2 week scan, 6 months post discharge
  The difference in quality of life outcomes (Medical Outcomes Study: 36-Item Short Form Survey) at 6 months post-hospital discharge between two groups randomized to undergo either a suprapatellar or infrapatellar approach to tibial IM nailing.
SMFA | Pre-op, 2 week scan, 6 months post discharge
  MFA46A Injury and Arthritis Survey

CONTACTS AND LOCATIONS:
Overall Officials: Samir Mehta, MD, Principal Investigator — University of Pennsylvania; Derek Donegan, MD, Principal Investigator — University of Pennsylvania; Annamarie Horan, PhD, Study Director — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States